CLINICAL TRIAL: NCT04113226
Title: Assessment of Survival and Autonomy With Rituximab Plus Chemotherapy or Rituximab Plus Lenalidomide for Elderly Patients With Relapsed Diffuse Large B-cell Lymphoma
Acronym: Relyage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: cimiez hospital Nice (Unknown); Institut Bergonié (Other); groupe hospitalier public sud de l'oise (Unknown); Henri Mondor University Hospital (Other); Centre Henri Becquerel (Other); Hôpital Charles Foix (Other); Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2018_843_0051
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Chemotherapy; Diffuse Large B-Cell Lymphoma (DLBCL), Nos; Elderly
Keywords: chemotherapy; Diffuse large B cell lymphoma (DLBCL); Relapse; activities of patients daily living; Elderly; Lenalidomide
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — Rituximab; Lenalidomide; Geriatric Assessment; Activities of Daily Living; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical rituximab-based chemotherapy (Active Comparator): Rituximab-based physician's choice chemotherapy
  Interventions: Drug: Rituximab; Other: Comprehensive Geriatric Assessment (CGA); Other: Activities of daily living (ADL) scale
- rituximab plus lenalidomide (Experimental): Four 28-days cycles of oral Lenalidomide (20 mg / d for 21 days) and Rituximab 375mg/m2 on day 1 and day 21. After this induction phase, patients achieving at least stable disease were given lenalidomide maintenance therapy (20 mg for 21 days) until progression.
  Interventions: Drug: Rituximab; Drug: Lenalidomide 20 MG; Other: Comprehensive Geriatric Assessment (CGA); Other: Activities of daily living (ADL) scale

INTERVENTIONS:
Drug: Rituximab — patients ≥ 75 years old with relapsed Diffuse large B-cell lymphoma will be treated with classical Rituximab-based chemotherapy or Rituximab plus Lenalidomide.
Drug: Lenalidomide 20 MG — patients ≥ 75 years old with relapsed Diffuse large B-cell lymphoma will be treated with Rituximab plus Lenalidomide. Four 28-days cycles of oral Lenalidomide (20 mg / d for 21 days) and Rituximab 375mg/m2 on day 1 and day 21. After this induction phase, patients achieving at least stable disease were given lenalidomide maintenance therapy (20 mg for 21 days) until progression
  Arms: rituximab plus lenalidomide
Other: Comprehensive Geriatric Assessment (CGA) — A comprehensive geriatric assessment (CGA) is recommended by the Société Internationale d'Onco Gériatrie (SIOG) in order to assess all geriatric facets (comorbidity, functional impairment, nutritional status, mental and psychological status, environment,…) on which treatment may impact.
Other: Activities of daily living (ADL) scale — Activities of daily living (ADL) comprise the basic actions that involve caring for one's self and body, including personal care, mobility, and eating. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.

SUMMARY:
Diffuse large B-cell lymphoma (DLBCL) is the most common type of non-Hodgkin lymphoma. Annual incidence increases with age and achieves more than 30 per 100 000 patients 65 years old or over.

Despite high response rates with conventional regimen as R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone), 30% to 40% of patients develop a relapse or a refractory disease, with a poor prognosis. There is no standard chemotherapy in second line for elderly patients, which are not eligible to receive a salvage treatment by high-dose therapy followed by autologous stem cell transplantation. The median progression-free-survival (PFS) is less than one year with the most commonly used regimens including R-Gemcitabine-Oxaliplatin (R-GEMOX) and R-Bendamustine. One the other side, Rituximab plus Lenalidomide, an immunomodulatory agent, is an active new therapeutic approach, with an efficacy proved in a phase II trial with a patients with a prolonged disease-free-survival of 32 months for responders in patients with a median age of 74 years old. This combination is also efficient in the ABC phenotype DLBCL which is more common in elderly patients.

For elderly patients, a management of the geriatric impairment together with lymphoma is required. Indeed, a comprehensive geriatric assessment detects frailty and vulnerability in elderly with a lymphoma and predicts severe treatment related toxicity, treatment settings and progression free survival. Moreover, geriatric intervention improved outcome, autonomy and quality of life. Functional status, assessed by Activities of patients Daily Living (ADL) is an independent predictive factor for feasibility of chemotherapy in elderly patients with cancer. The mini Data Set of DIALOG group is a new simplified geriatric assessment for oncologist.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years old
* Histologically proven CD20+ diffuse large B-cell lymphoma (DLBCL) (WHO classification 2008) including all clinical subtypes (primary mediastinal, intravascular, etc...), with all aaIPI. May also be included : transformed DLBCL from low grade lymphoma (Follicular, other...) and DLBCL associated with some small cell Infiltration in bone marrow or lymph node or CD20+ B-cell lymphoma, with intermediate features between DLBCL and Burkitt or with intermediate features between DLBCL and classical Hodgkin lymphoma or CD20+ Follicular lymphoma grade 3B or CD20+ Aggressive B-cell lymphoma unclassifiable
* Relapse ≥ 6 months
* ADL ≥ 2
* Negative HIV, HBV (anti-HBc negativity) and HCV serologies test within 4 weeks before inclusion
* Patient able to give his consent and having signed a written informed consent
* Registration in a national health-care system

Exclusion Criteria:

* Central nervous system or meningeal involvement by lymphoma
* Poor renal function (creatinine clearance < 30 ml/min, according to MDRD formula)
* Poor hepatic function (total bilirubin level>30mmol/l, transaminases >2.5 maximum normal level) unless these abnormalities are related to the lymphoma
* Neuropathy grade > 1
* Poor bone marrow reserve as defined by neutrophils<1.5 G/l or platelets<100 G/l, unless related to bone marrow infiltration
* Other concomitant or previous malignancy, except adequately treated in situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, or cancer in complete remission for <5 years
* Other serious and uncontrolled non-malignant disease.
* Insufficient proficiency of the French language and disability to complete a questionnaire
* Patient under guardianship

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression of free survival at 6 months in elderly patients treated with Rituximab plus Lenalidomide or Rituximab plus chemotherapy. | at 6 months
  Progression of free survival at 6 months with maintain autonomy without loss of 0.5 point of ADL in elderly patients 75 years old and over with relapsed diffuse large B-cell lymphoma treated with Rituximab plus Lenalidomide or Rituximab plus investigator's choice .

SECONDARY OUTCOMES:
Response rate in Rituximab plus Lenalidomide and Rituximab plus chemotherapy groups | at 6 months
  Response rate in Rituximab plus Lenalidomide and Rituximab plus chemotherapy groups
Overall survival rate in Rituximab plus Lenalidomide and Rituximab plus chemotherapy groups | at 6 months
  Response rate in Rituximab plus Lenalidomide and Rituximab plus chemotherapy groups

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Peyrade, MD, Principal Investigator — Centre Antoine Lacassagne, Nice; Boulhassass, MD, Principal Investigator — Hopital Cimiez NICE; Soubeyran, Pr, Principal Investigator — Institut Bergonié Bordeaux; Philippe Caillet, MD, Principal Investigator — Hôpital Henri Mondor, APHP CRETEIL; Fabrice Jardin, MD, Principal Investigator — Centre Henri Becquerel, ROUEN; Pascal Chaibi, MD, Principal Investigator — Hôpital Charles Foix, APHP IVRY/SEINE; Catherine Thieblemont, MD, Principal Investigator — Hôpital Saint-louis, APHP, PARIS; Damaj, MD, Principal Investigator — Centre Hospitalier Universitaire Caen; Garidi, MD, Principal Investigator — Centre Hospitalier SAINT-QUENTIN; Leduc, MD, Principal Investigator — Centre Hospitalier Abbeville; Dennetière, MD, Principal Investigator — Centre Hospitalier COMPIEGNE; Ivanoff, MD, Principal Investigator — Hôpital Avicenne, APHP BOBIGNY; Isabelle Grulois, MD, Principal Investigator — CH Saint Malo; Margot Robles, MD, Principal Investigator — CH Périgueux; Caroline DELETTE, PhD, Principal Investigator — CHU Amiens Picardie
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No